CLINICAL TRIAL: NCT01461356
Title: Prospective, Randomized, Controlled, Blinded Functional Outcomes Of Two Contemporary Surgical Approaches In Total Knee Arthroplasty
Brief Title: Minimally Invasive Surgical Approaches In Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Pagnano, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-001613
Record Dates: First submitted 2011-10-20; First posted 2011-10-28 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally Invasive Surgical approach (Experimental): Minimally invasive surgical approach for total knee replacement.
  Interventions: Procedure: Minimally invasive total knee replacement
- Medial Parapatellar surgical approach (Active Comparator): Standard medial parapateller surgical approach for total knee replacement.
  Interventions: Procedure: Standard approach total knee replacement

INTERVENTIONS:
Procedure: Minimally invasive total knee replacement — A cemented tricompartmental total knee replacement will be performed using a minimally invasive surgical approach.
  Other Names: Posterior stabilzed total knee replacement.; Minimally invasive total knee replacement.
  Arms: Minimally Invasive Surgical approach
Procedure: Standard approach total knee replacement — A cemented tricompartmental total knee replacement will be performed using a traditional medial parapatellar surgical approach.
  Other Names: Posterior stabilized total knee replacement.; Minimally invasive total knee replacment.
  Arms: Medial Parapatellar surgical approach

SUMMARY:
The hypothesis of the proposed study is that performing total knee arthroplasty through a mini subvastus approach results in statistically significant differences in one or more of the above functional outcome measures, when compared in a blinded, prospective, controlled, randomized manner to mini-medial arthrotomy approach.

1. Analyses of lower extremity functional activities (gait and stairs)
2. Strength of thigh musculature
3. Self-assessment of the functional outcomes
4. Return to the activities of daily living and sports activities

DETAILED DESCRIPTION:
In order to assign patients to specific treatment groups in an unbiased manner, randomization will occur prior to surgery. The assigned treatment codes for patients in each group will be generated by a computerized randomization program developed by the department of biostatistics, taking into account factors such age, sex and BMI. After the patient has met the entrance criteria, and given their full informed consent to participate in the study, they will be randomly assigned to one treatment group. Patient randomization will be performed during the clinic visit at which the surgery is scheduled, which typically occurs 1-3 days prior to surgery. The patients enrolled in the functional recovery measurement subset will be a consecutive series of the randomly assigned patients until 20 patients are assigned in each of the two study arms.

Operative Procedures The mini-subvastus approach and the medial parapatellar approach are the two surgical approaches that will be studied with respect to gait analysis, activity level and thigh strength. A cemented condylar implant, FDA approved devices, will be used for all cases in this study. The only difference between the two treatment groups will be the surgical approach for inserting these components. These two surgical approaches comprise the two study arms and are described in detail below.

Minisubvastus approach :

The skin incision is made from the superior pole of the patella to the top of the tibial tubercle and typically measures 3.5 inches in extension. The MIS subvastus approach is amenable to stepwise surgeon learning, and it is recommended that surgeons start with a traditional 6- to 8-in incision and then shorten the incision length as they gain familiarity with the subvastus exposure. The medial skin flap is elevated to clearly delineate the inferior border of the vastus medialis obliquus (VMO) muscle. The inferior border of the VMO is almost always found more inferior and more medial than most surgeons anticipate. This anatomy is very consistent, and the tendon at the inferior edge of the VMO attaches at a 50 degrees angle and attaches to the midpole of the patella. It is very important to save this edge of tendon as that is where the retractor will rest so that the VMO muscle itself is protected throughout the case. Incise with cautery along the inferior edge of the VMO over to the midpole of the patella (do not be tempted to cheat this superiorly as that will hinder, not help, the ultimate exposure). The proximal limb of the incision, which parallels the inferior edge of the VMO, is made at a 508 angle relative to the long axis of the femur. After intersecting the midpole of the patella the incision is directed straight distally along the medial border of the patellar tendon down to the inferior border of the tibial tubercle. A narrow 90 degrees bent Homan retractor is placed in the lateral gutter and rests against the robust edge of VMO tendon that was preserved during the exposure. The patella is completely retracted, with surprisingly little force, into the lateral gutter. The knee is then flexed to 90 degrees providing excellent exposure of the distal femur. If the patella does not slide easily into the lateral gutter with this maneuver it is typically because a portion of the medial patellofemoral ligament remains attached to the patella usually because the proximal limb of the arthrotomy was made in too horizontal a fashion rather than at the 50 degrees angle that parallels the VMO. The distal femur is prepared with a narrow version of a standard intramedullary resection guide. By bringing the knee out to 60 degrees of flexion the anterior portion of the distal femur can be visualized well. This position also relaxes the skin over the anterior femur making it easier to retract. If a very small skin incision is to be used, then the distal femur is cut one condyle at a time with the intramedullary portion of the cutting guide left in place for added stability. If a slightly longer skin incision is used, the distal cutting guide can be pinned in place and both condyles cut in a standard fashion. The tibia is prepared next and that is done to provide more working room for subsequently sizing and rotating the femoral component (the most difficult part of any MIS TKA). Good exposure of the entire surface of the tibia is accomplished with 3 retractors placed precisely: a pickle-fork retractor posteriorly to provide an anterior drawer and bent Homan retractors medially and laterally to protect the collaterals and define the perimeter of the tibial bone. The tibial resection is carried out with an extramedullary guide that is positioned under the skin but on top of the patellar tendon anteriorly. Because of this positioning, care must be taken to protect the patellar tendon during proximal tibial resection. The tibia is cut in one piece using a narrow but thick saw blade that fits the captured guide. The narrow blade allows sufficient maneuverability to work around the patellar tendon and sufficient tactile feedback for the surgeon to sense when the posterior and lateral tibial cortex has been cut. The femoral sizing and rotation guide is designed to be pinned to the distal femur and is thin enough that the knee can subsequently be brought out to 60 degrees of flexion to visualize the anterior femur for accurate sizing. By bringing the knee to 60 degrees of flexion and placing a retractor anteriorly the surgeon can confirm that the femoral cortex will not be notched. It is appropriate to clear some of the synovium overlying the anterior femoral cortex to be sure that femoral sizing is accurate and that the femur is not going to be notched. The femoral finishing guide can be translated medially or laterally and femoral rotation can be confirmed by referencing the posterior condyles, Whiteside's line, or the transepicondylar axis, all of which can be clearly defined with this subvastus approach. Before cutting the anterior femoral cortex the surgeon should confirm that the guide is placed appropriately to avoid notching. Trial components can be assembled and the knee reduced with a trial tibial insert to check overall limb alignment and flexion/ extension gap balance. Patellar preparation with this surgical approach can be saved until the end. Cutting the patella is not required for exposure, and by leaving the patella until the end the risk of inadvertent damage to the cut surface of the patella is minimized. The patella can be prepared freehand or with the surgeon's choice of cutting or reaming guides. If a cutting guide is used it is useful to remove the trial components before patellar preparation as then the entire limb can shorten, taking tension off the extensor mechanism and allowing easier access to the patella for preparation. The modular tibial tray is cemented first followed by the femur and then the patella. The tibia is subluxed forward with the aid of the pickle-fork retractor and the medial and lateral margins of the tibia are exposed well with 90 degrees bent Homan retractors. Care is taken to remove excess cement from around the tibial base plate, particularly posterolaterally, before moving on to cementing of the femur. The tibia is then repositioned under the femur at 90 degrees of flexion and the femur is exposed for cementing by placing bent Homan retractors on the medial and lateral sides above the collateral ligament insertions on the femur. A third retractor is placed under the VMO where it overlies the anterior femur. Cement is applied to both the posterior femoral condyles and the anterior femoral flange of the femoral implant and then cement is applied directly to the bone of the distal femur and anterior chamfer cuts. Alternately, the entire undersurface of femoral implant can be coated with cement before impaction. Care is again taken to remove all excess cement with special attention paid to the distal lateral surface of the femur where cement can extrude and be difficult to visualize once the patella is cemented. At this point the real tibial insert can be placed or a trial insert can be used as the surgeon sees fit. The patella is cemented last. Once the cement has hardened, patellar tracking is readily assessed. One should see centrally tracking without tilt or subluxation and contact of the patellar component with the medial femoral condyle with the knee in 908 of flexion. The tourniquet should be let down and any small bleeders in the subvastus space should be cauterized. The closure is begun by first reap proximating the corner of capsule at the midpole of the patella. Then, 3 interrupted 0-vicryl sutures are placed along the proximal limb of the arthrotomy. Care is taken to place those sutures deep to the VMO muscle itself and instead to grasp the underlying synovium attached to the VMO instead of the muscle itself. These first 4 sutures are then tied with the knee at 90 degrees of flexion to avoid oversewing the medial side and creating an iatrogenic patella baja postoperatively. A deep drain is placed in the knee joint and the distal/vertical limb of the arthrotomy is closed with multiple interrupted 0-vicryl sutures placed with the knee in 90 degrees of flexion. The skin is closed in layers. Staples are preferred over a subcuticular suture for the final closure. There is unquestionably more tension placed on the skin during any MIS TKA surgery than is the case in standard open surgery and, in our experience, the potential for wound healing problems is magnified if the skin is handled multiple times as is the case with a running subcuticular closure.

Standard Approach:

A medial parapatellar approach will be performed in the control group; this is a contemporary modification to the standard approach for total knee arthroplasty.

Postoperative Course Hospitalization Patients will come into the hospital on the day of their surgery. Hospitalization of 2 to 3 nights is routine for these patients, although complications may prolong that time. The patient will receive one preoperative dose and three postoperative doses of IV antibiotics over a 24 hour period. All patients will receive appropriate anticoagulation for deep venous thrombosis prophylaxis.

Postoperative Physical Therapy

Both treatment groups will have identical postoperative care via standard postoperative clinical pathways. Structured physical therapy will begin the day after surgery and continued during the hospitalization. Patients are encouraged to sit up at the bedside the evening of their surgery. A home therapy program will be given to the patient, although formal physical therapy will not continue on an outpatient basis. The following general principles will be followed and the patient instructed accordingly:

* Post-op Day 1, transfer from bed to chair with assist
* Active ROM to begin within first 24 hours postoperatively
* Weight bearing status and progression as tolerated
* Progress ambulation from walker to crutches/cane(s) as tolerated
* Patients should be encouraged to maximize independent ambulation and increase distance ambulated daily

Discharge Criteria

* Patient is independent and safe with aids
* Patient is able to transfer out of and into bed from a standing position
* Is able to rise from a chair to a standing position
* Ambulate 100 feet

ELIGIBILITY:
Inclusion Criteria:

* Primary arthroplasty
* Age between 45 and 75 years old
* Single condylar implant design

Exclusion Criteria:

* Revision arthroplasty
* Age less than 45 and greater than 75 years old
* Pre-operative flexion lower than 90 degrees
* Valgus or varus knee deformity greater than 15 degrees.
* The presence of infections, highly communicable diseases (AIDS, active tuberculosis, venereal disease, hepatitis) or metastasis disease.
* Significant neurological or musculoskeletal disorders or disease that may interfere with normal gait or weight bearing.
* Any congenital, developmental, or other bone disease or previous hip surgery that may, in the surgeon's judgment, interfere with TK prosthesis survival or success.
* Presence of previous prosthetic knee or hip replacement device.
* BMI > 30.
* Pregnant women.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Knee Society Clinical Rating Score | 2 months
  The two patient cohorts, minimally invasive surgical approach and standard medial parapatellar approach, will be followed prospectively and evaluated with the Knee Society Clinical Rating Score.

SECONDARY OUTCOMES:
Comprehensive gait analysis | 2 months
  Spatiotemporal gait parameters will be measured in the gait analysis lab and compared between the two groups to determine if a functional difference is detectable between the two different surgical approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Pagnano, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States